CLINICAL TRIAL: NCT04482673
Title: The Role of Vitamin D in Mitigating COVID-19 Infection Severity: Focusing on Reducing Health Disparities in South Carolina
Brief Title: Vitamin D Supplementation in the Prevention and Mitigation of COVID-19 Infection
Acronym: VitD-COVID19
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Grassroots Health Nutrition Institute (Unknown); ZRT Laboratory (Other)
Responsible Party: Principal Investigator, Carol L. Wagner, MD, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00099939
Record Dates: First submitted 2020-07-01; First posted 2020-07-22 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Vitamin D Deficiency; Respiratory Viral Infection
Keywords: COVID-19; Vitamin D Deficiency; Respiratory Viral Infection
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- COVID-19 Negative Active Treatment (Experimental): Participants will be randomized to vitamin D3 (6000 IU) per day for 12 months. All participants will receive a multivitamin containing 800 IU vitamin D3/day.
  Interventions: Drug: Daily Vitamin D3
- COVID-19 Negative Placebo (Placebo Comparator): Participants in this arm would receive placebo for 12 months. All participants will receive a multivitamin containing 800 IU vitamin D3/day.
  Interventions: Drug: Daily placebo
- COVID-19 Positive Active Treatment (Experimental): Participants will be randomized to vitamin D3 as a bolus (20,000 IU) per day for 3 days followed by high dose vitamin D (6000 IU) per dayfor 12 months. All participants will receive a multivitamin containing 800 IU vitamin D3/day.
  Interventions: Drug: Daily Vitamin D3; Drug: Bolus vitamin D3
- COVID-19 Positive Placebo (Placebo Comparator): Participants in this arm would receive placebo as a bolus followed by daily placebo for 12 months. All participants will receive a multivitamin containing 800 IU vitamin D3/day.
  Interventions: Drug: Daily placebo; Drug: Bolus placebo

INTERVENTIONS:
Drug: Daily Vitamin D3 — 6000 IU vitamin D3 daily
  Other Names: Daily cholecalciferol
  Arms: COVID-19 Negative Active Treatment; COVID-19 Positive Active Treatment
Drug: Daily placebo — Placebo daily
  Arms: COVID-19 Negative Placebo; COVID-19 Positive Placebo
Drug: Bolus vitamin D3 — Bolus 20,000 IU vitamin D3 daily for 3 days
  Other Names: Bolus cholecalciferol
  Arms: COVID-19 Positive Active Treatment
Drug: Bolus placebo — Bolus placebo daily for 3 days
  Arms: COVID-19 Positive Placebo

SUMMARY:
The purpose of this study is to evaluate how useful vitamin D supplementation is in reducing the severity of COVID-19 symptoms and the body's inflammatory and infection-fighting response to COVID-19. Individuals ≥50 years of age and older who are tested for COVID-19 and negative will be randomized (like flipping a coin) to either daily high dose vitamin D supplementation (6000 IU vitamin D3/day) vs. standard of care. Those individuals ≥50 years of age or older who test positive for COVID-19 at baseline will be randomized to bolus vitamin D (20,000 IU/day for 3 days) followed by high dose (6000 IU vitamin D/day) vs. standard of care for 12 months. All participants will receive a multivitamin containing vitamin D.

DETAILED DESCRIPTION:
Vitamin D (vitD) deficiency is more prevalent among African Americans and Latinx and in the elderly who have low exposure to sunlight. African Americans and nursing home residents who contract SARS-CoV-2, the novel virus that first appeared in Wuhan, China, and who develop the disease designated COVID-19 experience a much worse clinical outcome than other groups. Some have speculated that low vitD status could exacerbate COVID-19 infection, especially if the viral infection reaches the lower respiratory tract.

Sufficient vitD may help to improve the pulmonary immune response to the virus, reduce the dangerous cytokine storm, and lessen surfactant dysregulation, potentially preventing or ameliorating the acute syndrome. To maximize the benefits of vitD on host response to SARS-CoV-2, prophylactic supplementation to ensure sufficiency before COVID-19 would be the preferable public health option. Yet, vitD supplementation during acute infection may also improve overall clinical outcome in some infected patients. It is a relatively inexpensive therapy that has a large safety profile when given in doses of 4000-6000 international units/day to adults.

To date, there is no effective cure or preventive vaccine for COVID-19. Given the risk of disease and death, any intervention that reduces the morbidity and mortality from COVID-19 would be of immense value. We hypothesize that achieving and sustaining vitD sufficiency through dietary supplementation will result in improved immune function and a decrease in COVID-19 incidence and symptomatology. Importantly, this objective will address the significant health disparity of vitD deficiency among black, Latina and the elderly. We further hypothesize that those individuals with a circulating 25(OH)D of ≥40 ng/mL will have less severe COVID-19 symptoms, particularly among higher risk populations. We will compare the effectiveness of higher dose vitD vs. standard of care dosing.To test these hypotheses, we propose the following Aims:

1. Focusing on prevention, this Aim will test whether achieving vitD sufficiency (as defined by total circulating 25(OH)D ≥40-60 ng/mL) in individuals at risk for deficiency will improve clinical outcomes in those who subsequently develop COVID-19.
2. Focusing on vitD as mitigation therapy, this Aim will evaluate the effectiveness of bolus dosing followed by daily vitD supplementation in achieving the target 25(OH)D range of ≥40-60 ng/mL in those individuals testing positive for COVID-19 at MUSC/affiliated hospital facilities, but do not require admission to a hospital (outpatient) and will examine whether achieving this target range is associated with less severe COVID-19 and differences in inflammatory cytokine profiles.

In the prevention arm of this project (Aim 1), individuals at higher risk ≥50 years of age who test negative for COVID-19 at MUSC/its affiliate hospitals, and agree to daily vitD supplementation for a 12-month period, with vitD status measured monthly will be randomized to placebo or prescribed vitD (6000 IU/day) to achieve a total circulating 25(OH) concentration of ≥40-60 ng/mL. We will compare study groups regarding subsequent infection with COVID-19, severity of symptoms, need and duration of hospitalization (LOS), admission to the ICU, need for ventilatory support, and mortality, along with return to baseline activities and/or work, as a function of age, BMI, and other recognized COVID-19 risk factors. In the mitigation arm of this project (Aim 2), non-hospitalized individuals ≥50 years of age who test COVID-19 positive will be randomized to placebo or a bolus of oral vitD (20,000 IU X 3 days) followed by 6000 IU vitD/day, and we will compare study groups on measures of disease severity as in Aim 1. All participants in both Aims 1 and 2 will receive a daily multivitamin (MVI) containing 800 IU VitD for the 12-month period.

Following the completion of these Aims, we will be able to answer the following questions:

1. Are individuals with vitD deficiency more likely to be diagnosed with COVID-19 infection?
2. Does being vitD replete make a person more likely to have asymptomatic COVID-19?
3. Does vitD sufficiency status account for why African Americans, Latina, and the elderly more likely to experience complications related to COVID-19?
4. Is vitD deficiency in COVID-19 positive outpatients associated with increased severity of symptoms and differences in inflammatory cytokine profiles that is mitigated by bolus and then sustained vitD supplementation?

The long-term impact of these studies will influence public policy regarding more widespread vitD supplementation is a means of reducing the severity of COVID-19. Given its low cost and the ease with which widespread supplementation could be instituted, oral vitD supplementation may represent a rapid and inexpensive means by which to reduce both the COVID-19 incidence and severity.

ELIGIBILITY:
Entry Criteria:

---Adults aged 50 years of age or older who presents to MUSC or its affiliate hospitals (or associated testing centers) for COVID-19 testing during the recruitment period is eligible for participation.

Exclusion Criteria:

* Hospitalization at the time of study recruitment.
* Any individual less than 50 years of age. The reason that the participants ≥50 years are being excluded from this study is because those who are ≥50 years have a higher risk of being symptomatic with COVID-19 and have the potential for the greatest benefit. The disease appears to manifest differently in children and its occurrence is quite rare.
* Only those patients tested for COVID-19 initially will be eligible to participate; therefore, anyone wanting to participate in the trial must have had a COVID-19 test prior to enrollment/participation in the study.
* Any individual who is not capable of making independent decisions and who is considered cognitively impaired.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in total circulating 25(OH)D concentration | monthly in COVID-19 negative participants through study completion for 1 year
  metabolite of vitamin D
Change in total circulating 25(OH)D concentration in COVID-19 positives | baseline, 2 and 4 weeks, then months 3, 6, 9 and 12 in COVID-19 positive participants
  metabolite of vitamin D
Change in SARS-CoV-2 antibody titers | every 3 months up to 12 months
  The presence or absent of SARS-CoV-2 antibody will be measured at baseline, 3, 6, 9 and 12 months.

SECONDARY OUTCOMES:
Change in inflammatory cytokine concentration (10 cytokine panel Elisa: Interferon (INF)-gamma, Interleukin (IL)-1beta, IL-2, IL-3, IL-4, IL-6, IL-8, IL-10, IL-13, Tumor Necrosis Factor (TNF)-alpha | baseline and every 3 months up to 12 months
  At baseline, 3, 6, 9 and 12 months, inflammatory cytokines will be measured in participant plasma samples. Cytokines to be measured are Interferon-gamma (IFN-g), Interleukin-1beta (IL-1B), IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-13, and Tumor Necrosis Factor-alpha (TNFa). Values of these cytokines at baseline will compared to those at 3, 6, 9, and 12 months
Respiratory symptoms | daily for 2 weeks
  COVID-19 positive participants or if COVID-19 negatives develop respiratory symptoms will complete this respiratory survey daily for 2 weeks
Signs and symptoms of rhino/sinusitis | Baseline then 3, 6, 9 and 12 months in negatives and daily for 2 weeks in positives
  Inventory of signs and symptoms of rhino/sinusitis. These signs include sneezing, running nose, cough, dizziness, fatigue, and sense of smell. Each sign is rated on a scale of 0 to 5, with 0 indicating not problem, for instance 1 indicating mild problem, 4 indicating severe problem and 5 indicating problem as bad as it can be.
NCI Dietary Intake | baseline then at 6 and 12 months
  Dietary intake assessment
Charlson Comorbidity survey | baseline then at 6 and 12 months
  Survey of participant health problems
Paffenberger Physical Activity Assessment | Baseline then at 6 and 12 months
  Assessment of physical activity of each participant
Perceived stress | monthly for 1 year
  Each participant will complete the Perceived Stress Scale Questionnaire (PSS) to assess their perceived stress. Assessments are base on a scale of 0 to 4, with 0 indicating "never" and 4 indicating "very often"
Pandemic stress | monthly for 1 year
  Each participant will complete the and Pandemic Stress Index Questionnaire (PSI) to assess their perceived stress cause by the pandemic. Assessments are base on a scale of 0 to 6, with 0 indicating "not at all" and 5 indicating "extremely," and 6 indicating "decline to answer."
NEO-Personality Inventory | baseline visit
  Personality characteristics of each participant
GrassrootsHealth Monthly Health assessment | baseline, 6, and 12 months
  A health assessment will be completed by each participant monthly for 1year. This health. This is for information on health status only and not for comparative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Wagner, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No